CLINICAL TRIAL: NCT05897710
Title: Virtual World-Based Cardiac Rehabilitation to Improve Cardiovascular Health and Outcomes Among Cardiac Patients
Brief Title: Virtual World-Based Cardiac Rehabilitation
Acronym: VWCR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Johns Hopkins University (Other); University of California, Irvine (Other); University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, LaPrincess C. Brewer, Associate Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-011357
Record Dates: First submitted 2023-05-05; First posted 2023-06-09 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Cardiac Event; Telemedicine; Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Center-Based Cardiac Rehab (CBCR) (Active Comparator): Standard of care for participants' center-based cardiac rehabilitation program. Traditional 12-week, in-person program.
  Interventions: Other: Center-Based Cardiac Rehabilitation (CBCR)
- Virtual World-Based Cardiac Rehab (VWCR) (Experimental): Telehealth delivery of cardiac rehabilitation via Second Life virtual world platform. 12-week, home-based program.
  Interventions: Other: Virtual World-Based Cardiac Rehabilitation (VWCR)

INTERVENTIONS:
Other: Virtual World-Based Cardiac Rehabilitation (VWCR) — 12-week virtual world technology-based program via Second Life platform. Weekly virtual visits with nurse coach and exercise physiologist, weekly education sessions, and social support group discussions within the virtual world environment.
  Other Names: Destination Cardiac Rehab
  Arms: Virtual World-Based Cardiac Rehab (VWCR)
Other: Center-Based Cardiac Rehabilitation (CBCR) — Traditional 12-week in-person cardiac rehabilitation program; standard of care at participant's cardiac rehabilitation facility
  Arms: Center-Based Cardiac Rehab (CBCR)

SUMMARY:
The proposed trial is a multiphase, multicenter, non-inferiority, hybrid type 1 effectiveness, randomized controlled trial to test an innovative virtual world-based cardiac rehabilitation (CR) program, "Destination Cardiac Rehab". The primary objectives of this study are to assess the efficacy and adherence of "Destination Cardiac Rehab" compared to traditional center-based CR.

DETAILED DESCRIPTION:
The proposed virtual world-based cardiac rehabilitation (VWCR) program provides a novel home-based delivery method of a CR program to address several barriers to care associated with traditional center-based CR (CBCR). This 2-arm, randomized controlled trial (RCT) will rigorously assess adherence and efficacy of VWCR compared to CBCR in a 12-week (36-session) intervention that includes patient education, self-monitoring of physical activity and blood pressure, social support, and weekly telehealth visits with a CR nurse and exercise physiologist. Patients with a CR eligible cardiovascular event will be recruited from 6 geographically diverse CR centers across the United States. We hypothesize that the VWCR, known as "Destination Cardiac Rehab" will be non-inferior to CBCR as assessed by improvement in cardiovascular health and adherence to CR sessions.

ELIGIBILITY:
Inclusion Criteria:

* Indication for CR according to Centers for Medicare & Medicaid Services (CMS) guidelines: Myocardial infarction within the preceding 12 months; Coronary artery bypass surgery; Current stable angina (chest pain); Heart valve repair or replacement; Percutaneous transluminal coronary angioplasty (PTCA) or coronary stenting; Heart or heart-lung transplant; Stable chronic heart failure
* Aged ≥18 years
* Basic Internet navigation skills
* Active email address

Exclusion Criteria:

* High risk patients according to the American Association of Cardiovascular and Pulmonary Rehabilitation (AACVPR) risk stratification (e.g., sudden cardiac arrest survivor)
* Receiving continuous inotropic support
* Presence of a mechanical circulatory support device
* Decompensated heart failure
* Symptomatic valvular heart disease
* Uncontrolled angina
* Presence of hemodynamically unstable dysrhythmias (e.g., ventricular tachycardia) given safety concern of unsupervised exercise20
* Pregnant (due to associated hormonal and weight changes)
* Non-English-speaking
* Visual/hearing impairment or mental disability that would preclude independent use of the VW platform

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2881 (Actual)
Dates: Start 2023-03-07 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Life's Essential 8 component: Self-reported healthy diet | Baseline, 3 months, and 6 months post-randomization
  Changes from baseline in healthy diet using the Mediterranean Eating Patterns for Americans (MEPA), a 16-item questionnaire evaluating accordance with a Mediterranean-like diet pattern
Life's Essential 8 component: Self-reported physical activity | Baseline, 3 months, and 6 months post-randomization
  Changes from baseline in physical activity using the International Physical Activity Questionnaire (IPAQ), a 12-item questionnaire classifying physical activity as "low," "moderate," or "high" intensity physical activity (minutes/day) over the prior week
Life's Essential 8 component: Self-Reported smoking status | Baseline, 3 months, and 6 months post-randomization
  Changes from baseline in smoking status using the National Health and Nutrition Examination Survey-Smoking-Cigarette Use Questionnaire (NHANES-SMQ), evaluating current and past smoking habits
Life's Essential 8 component: Sleep Quality | Baseline, 3 months, and 6 months post-randomization
  Changes from baseline in sleep quality (number of hours of sleep nightly) using the Pittsburg Sleep Quality Index (PSQI).
Life's Essential 8 component: Body Mass Index (BMI) | Baseline, 3 months, and 6 months post-randomization
  Changes from baseline in BMI as calculated with weight (kg) and height (m), reported as kg/m^2
Life's Essential 8 component: Cholesterol | Baseline, 3 months, and 6 months post-randomization
  Changes from baseline in Non-HDL Cholesterol levels reported as mg/dL
Life's Essential 8 component: Blood Glucose | Baseline, 3 months, and 6 months post-randomization
  Changes from baseline in Hemoglobin A1c (percent) and fasting blood glucose (mg/dL)
Life's Essential 8 component: Blood Pressure | Baseline, 3 months, and 6 months post-randomization
  Changes from baseline in systolic and diastolic blood pressure measurements; average of three sitting readings in mmHg
Life's Essential 8 composite score: Cardiovascular health | Baseline, 3 months, and 6 months post-randomization
  Changes from baseline in Life's Essential 8 score. Life's Essential 8 composite score is determined as a composite of all components by calculating an unweighted average score on a scale of 0 to 100 points. An overall cardiovascular health score (Life's Essential 8 score) will be considered high (80 to 100 points), moderate (50 to 79 points) or low for (0 to 49 points).
Number of sessions attended by participants | Baseline through 12-week program
  Optimal adherence defined as completion of 70% or more of weekly visits (in-person or virtual). Attendance measured by CR staff for control group, and by VWCR web administrators, Exercise Physiologists, and Nurse Coaches in the VWCR arm.

SECONDARY OUTCOMES:
MACE (Major Adverse Cardiovascular Events) 3 months post-randomization | 3 months and 6 months post-randomization
  MACE (Major Adverse Cardiovascular Events): CV-related hospital readmissions; CV and all-cause mortality
Exercise Sessions | Baseline through 12-week (36 session) cardiac rehabilitation program
  Self-reported number of self-directed exercise sessions per week, confirmed by Fitbit activity tracker data.
Functional Capacity | Baseline, 3 months, and 6 months post-randomization
  Six-Minute walk test, evaluating blood pressure, oxygen saturation, and pulse after walking for 6 minutes at a normal pace
Health-related quality of life | Baseline, 3 months, and 6 months post-randomization
  Changes from baseline in health-related quality of life using the Short Form [SF]-12 Health Survey, a self-reported outcome measure assessing the impact of health on an individual's everyday life. The SF-12 consists of 12-items and 8 subdomains. Each item of the questionnaire has response categories which vary from 2- to 6-point scales and raw scores for items ranging from 1 to 6. The raw scores are summated and linearly transformed into 0-100 scale with a higher score indicating better health status.
Physical Activity Self-efficacy | Baseline, 3 months, and 6 months post-randomization
  Changes from baseline in physical activity self-efficacy measured by the Exercise Confidence Survey scale to assess the participant's confidence in their ability to exercise when faced with common barriers. 12 items are assessed, each on a 5-point scale ranging from 1 to 5. A higher total sum indicates higher self-efficacy for physical activity.
Physical Activity Self-regulation | Baseline, 3 months, and 6 months post-randomization
  Changes from baseline in physical activity self-regulation measured by the Health Beliefs Survey to assess strategies used in the past 3 months to increase their step count or physical activity levels. Items are measured on a five-point scale from 1 (never) to 5 (repeatedly). Higher scores indicate more self-regulation.
Physical Activity Social Support | Baseline, 3 months, and 6 months post-randomization
  Changes from baseline in physical activity social support using the Social Support for Exercise Survey scale that asks participants how much encouragement they received to increase physical activity on a five-point scale from 1 (never) to 5 (very often). Higher scores indicate more social support for physical activity.
Diet Self-efficacy | Baseline, 3 months, and 6 months post-randomization
  Changes from baseline in diet self-efficacy measured the Diet Confidence Survey scale to assess the participant's confidence in their ability to maintain a healthy diet when faced with common barriers. 12 items are assessed, each on a 5-point scale ranging from 1 to 5. A higher total sum indicates higher self-efficacy for healthy eating.
Diet Self-regulation | Baseline, 3 months, and 6 months post-randomization
  Changes from baseline in diet self-regulation measured by the Health Beliefs Survey to assess strategies used in the past 3 months to eat healthier foods. Items are measured on a five-point scale from 1 (never) to 5 (repeatedly). Higher scores indicate more use of self-regulation strategies to promote healthy eating.
Diet Social Support | Baseline, 3 months, and 6 months post-randomization
  Changes from baseline in diet social support using the Social Support for Eating Habits Survey scale that asks participants how much encouragement they received to eat healthier on a five-point scale from 1 (never) to 5 (very often). Higher scores indicate more social support for healthy eating.

CONTACTS AND LOCATIONS:
Overall Officials: LaPrincess Brewer, M.D., M.P.H., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brewer LC, Abraham H, Clark D 3rd, Echols M, Hall M, Hodgman K, Kaihoi B, Kopecky S, Krogman A, Leth S, Malik S, Marsteller J, Mathews L, Scales R, Schulte P, Shultz A, Taylor B, Thomas R, Wong N, Olson T. Efficacy and Adherence Rates of a Novel Community-Informed Virtual World-Based Cardiac Rehabilitation Program: Protocol for the Destination Cardiac Rehab Randomized Controlled Trial. J Am Heart Assoc. 2023 Dec 5;12(23):e030883. doi: 10.1161/JAHA.123.030883. Epub 2023 Nov 28. PMID 38014699